CLINICAL TRIAL: NCT05671393
Title: A Multi-institution Real-world Study of the Optimal Surveillance Frequency for Patients With Gastric Neuroendocrine Carcinoma
Brief Title: the Optimal Surveillance Frequency for Patients With Gastric Neuroendocrine Carcinoma
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director of gastric surgery, Fujian Medical University
Other Study IDs: FUNEC-01
Record Dates: First submitted 2022-12-31; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Gastric Neuroendocrine Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to lacking of evidence on surveillance for gastric neuroendocrine carcinoma (G-NEC), this study aimed to determine the optimal postsurgical surveillance strategy for G-NEC patients and compare its cost-effectiveness with traditional surveillance strategies.

DETAILED DESCRIPTION:
The development of existing follow-up strategies is mainly based on experts' consensus and researches on recurrence patterns due to the lack of direct evidence and unified standards. On the one hand, it is unreasonable to carry out the same postoperative surveillance for all G-NEC patients. In addition to the early detection of recurrence, the optimal follow-up strategy should also balance cost and effectiveness. There were no criteria for the arrangement of follow-up in different guidelines, and the optimal postoperative follow-up strategy for patients with G-NEC remains unclear. Patients with G-NEC from 21 centers in China were included. Cost-effectiveness were assessed by Markov model.

ELIGIBILITY:
Inclusion Criteria:This multicentre retrospective study included patients with gastric neuroendocrine neoplasms who underwent surgery in 21 centres of the Study Group for Gastric Neuroendocrine Tumours in China from January 2008 to December 2016. Radical surgery included a D2 lymphadenectomy consistent with the Japanese gastric cancer treatment guidelines.

Exclusion Criteria: Patients with tumours of unknown pathology (only neuroendocrine neoplasms recorded without detailed information); patients with gastric NETs; patients who had endoscopic submucosal dissection or endoscopic mucosal resection; patients who received neoadjuvant chemotherapy; patients who died within 3 months of surgery from postoperative complications; and patients with unknown tumour size or who were lost to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 801 G-NEC patients from 21 centers in China were included.
Sampling Method: Non-Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
recurrence rate | 60 months
  distant, peritoneal, and local recurrence

SECONDARY OUTCOMES:
Delayed-detection months | 60 months
  A hypothetical cohort of 1000 G-NEC patients was generated to compare the effectiveness of surveillance among the above-mentioned strategies by calculating the sum of the delayed detection months. Delayed detection months were defined as the duration from the occurrence of failure to the next-nearest follow-up. For instance, if a patient develops distant metastasis in the 3rd month while the next nearest planned visit is in the 5th month, the delayed -detection time for this patient is 2 months. The total number of delayed detection months of our risk-based surveillance schedule and that of the control strategies were simulated and compared.
Incremental cost-effectiveness ratios (ICERs) | 60 months
  ICERs were calculated by dividing the difference in cost by the difference in QALY

CONTACTS AND LOCATIONS:
Overall Officials: Chang-ming Huang, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Chang-ming Huang, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu BB, He XY, Zhou YB, He QL, Tian YT, Hao HK, Qiu XT, Jiang LX, Zhao G, Li Z, Xu YC, Fu WH, Xue FQ, Li SL, Xu ZK, Zhu ZG, Li Y, Li E, Chen JP, Li HL, Cai LS, Wu D, Li P, Zheng CH, Xie JW, Lu J, Huang CM. Optimal postoperative surveillance strategies for cancer survivors with gastric neuroendocrine carcinoma based on individual risk: a multicenter real-world cohort study. Int J Surg. 2023 Jun 1;109(6):1668-1676. doi: 10.1097/JS9.0000000000000401. PMID 37076132